CLINICAL TRIAL: NCT05400746
Title: A Phase Ia Study to Assess Safety and Immunogenicity of the Plasmodium Falciparum Malaria Vaccine Candidate Pfs48/45 in Matrix-M Adjuvant in Healthy Adults Living in the UK
Brief Title: A Study of the Plasmodium Falciparum Malaria Vaccine Candidate Pfs48/45 in Matrix-M Adjuvant in the UK
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Significant delays in vaccine adjuvant supply due to an out of specification within the context of the grant timeline. Limited safety and immunological data could be accrued from incomplete regimens.
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC085
Record Dates: First submitted 2022-05-26; First posted 2022-06-02 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2023-05

CONDITIONS: Malaria; Plasmodium Falciparum
Keywords: Pfs48/45; Matrix-M
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Matrix-M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - low dose (Experimental): 8-10 volunteers receiving three doses of 10 µg Pfs48/45 in 50 µg Matrix-M on days 0, 28 and 56 via intramuscular injection (IM) in the deltoid region of the arm
  Interventions: Biological: Pfs48/45 in Matrix-M
- Group 2 - standard dose (Experimental): 8-10 volunteers receiving three doses of 50 µg Pfs48/45 in 50 µg Matrix-M on days 0, 28 and 56 via intramuscular injection (IM) in the deltoid region of the arm
  Interventions: Biological: Pfs48/45 in Matrix-M
- Group 3 - fractional dose (Experimental): 8-10 volunteers receiving two doses of 50 µg Pfs48/45 in 50 µg Matrix-M on days 0 and 28, followed by one dose of 10 µg Pfs48/45 in 50 µg Matrix-M on day 56 via intramuscular injection (IM) in the deltoid region of the arm
  Interventions: Biological: Pfs48/45 in Matrix-M

INTERVENTIONS:
Biological: Pfs48/45 in Matrix-M — Three doses of Pfs48/45 in Matrix-M at different doses

SUMMARY:
This is an open label, single-site, first-in-human, dose-escalation Phase Ia study to assess safety and immunogenicity of the Plasmodium falciparum malaria vaccine candidate Pfs48/45 in Matrix-M adjuvant in healthy adults living in the UK

DETAILED DESCRIPTION:
Volunteers will be recruited into one of three groups (n=8-10 per group) at the Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford over approximately 12 months. All volunteers will receive three dose of Pfs48/45 in 50 µg Matrix-M, administered intramuscularly and given four weeks apart. Enrolment will be staggered with clinical and safety reviews, follow-up visits and monitoring via a diary card.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their GP.
* Volunteers with the potential to become pregnant only: must practice continuous effective contraception for the duration of the study (see section 10.10).
* Agreement to refrain from blood donation for the duration of the study.
* Able and willing to provide written informed consent to participate in the trial

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months.
* Use of immunoglobulins or blood products (e.g., blood transfusion) in the last three months.
* Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days following each study vaccination, with the exception of COVID-19 vaccines, which should not be received between 14 days before to 7 days after any study vaccination.
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Concurrent involvement in another clinical trial or planned involvement during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data, as assessed by the Investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any history of anaphylaxis in reaction to vaccinations.
* Pregnancy, lactation or intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 25 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless volunteer has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV ribonucleic acid (RNA) PCR at screening for this study).
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested. Procedures for identifying laboratory values meeting exclusion criteria are shown in SOP VC027.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Inability of the study team to contact the volunteer's GP to confirm medical history.

Absolute contraindications:

* Anaphylactic reaction following administration of vaccine.
* Pregnancy.

Contraindications at that point in time (may be rescheduled):

* Acute disease at the time of vaccination. (Acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e. temperature of ≤37.5°C/99.5°F.
* Temperature of >37.5°C (99.5°F) at the time of vaccination.
* Current COVID-19 infection, defined as ongoing symptoms with positive COVID-19 PCR swab test taken during current illness or positive COVID-19 PCR swab or rapid antigen test within preceding 7 days without symptoms. Vaccinations will be delayed by a minimum of 7 days from the date of the first positive COVID-19 PCR swab or rapid antigen test, as long as symptoms are improving or resolved. It will be at the discretion of the Investigator to withdraw a participant if they develop severe COVID-19 disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, DPhil FRCP, Principal Investigator — Center for Clinical Vaccinology and Tropical Medicine, University of Oxford
Locations (1):
- CCVTM, Churchill Hospital, University of Oxford, Oxford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose
Started | 8 | 8 | 1
Completed | 8 | 4 | 0
Not Completed | 0 | 4 | 1
Not completed — Trial terminated early due to IMP availability | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose | Total
Number analyzed (Participants) | 8 | 8 | 1 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 1 | 17
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 1 | 10
  Male | 5 | 2 | 0 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Other Asian background | 1 | 0 | 0 | 1
  White - British | 4 | 7 | 1 | 12
  White - Other | 2 | 0 | 0 | 2
  Asian or Asian British - Bangladeshi | 0 | 1 | 0 | 1
  Hispanic | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of the Pfs48/45 With Matrix-M Vaccine at Various Doses in Healthy Adult Volunteers by Assessing the Occurrence of Solicited Local Reactogenicity Signs and Symptoms for 7 Days Following Each Vaccination
Description: Occurrence of solicited local reactogenicity signs and symptoms for 7 days following each vaccination using e-diaries, clinical review, clinical examination (including observations) and laboratory results
Time Frame: 7 days following each vaccination
Measure: Number; unit: Number of participants reporting events
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose
Number analyzed (Participants) | 8 | 8 | 1
Number of participants reporting events
  Pain (Mild) | 7 | 6 | 0
  Pain (Moderate) | 2 | 3 | 0
  Pain (Severe) | 0 | 0 | 0
  Warmth (Mild) | 4 | 6 | 0
  Warmth (Moderate) | 1 | 0 | 0
  Warmth (Severe) | 0 | 0 | 0
  Itch (Mild) | 2 | 0 | 0
  Itch (Moderate) | 1 | 0 | 0
  Itch (Severe) | 0 | 0 | 0
  Redness | 7 | 5 | 1

2. Primary Outcome: Safety and Tolerability of the Pfs48/45 With Matrix-M Vaccine at Various Doses in Healthy Adult Volunteers by Assessing the Occurrence of Solicited Systemic Reactogenicity Signs and Symptoms for 7 Days Following Each Vaccination
Description: Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following each vaccination using e-diaries, clinical review, clinical examination (including observations) and laboratory results.
Time Frame: 7 days following each vaccination
Measure: Number; unit: Number of participants reporting events
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose
Number analyzed (Participants) | 8 | 8 | 1
Number of participants reporting events
  Arthralgia (mild) | 5 | 3 | 0
  Arthralgia (moderate) | 3 | 2 | 0
  Arthralgia (severe) | 0 | 0 | 0
  Myalgia (mild) | 5 | 5 | 0
  Myalgia (moderate) | 3 | 2 | 0
  Myalgia (severe) | 0 | 1 | 0
  Fever (mild) | 2 | 3 | 0
  Fever (moderate) | 3 | 2 | 0
  Fever (severe) | 0 | 0 | 0
  Headache (mild) | 6 | 7 | 1
  Headache (moderate) | 4 | 4 | 0
  Headache (severe) | 0 | 0 | 0
  Fatigue (mild) | 6 | 7 | 0
  Fatigue (moderate) | 2 | 3 | 0
  Fatigue (severe) | 1 | 0 | 0
  Nausea (mild) | 2 | 3 | 0
  Nausea (moderate) | 0 | 0 | 0
  Nausea (severe) | 0 | 0 | 0
  Malaise (mild) | 5 | 6 | 0
  Malaise (moderate) | 3 | 1 | 0
  Malaise (severe) | 0 | 0 | 0

3. Primary Outcome: Safety and Tolerability of the Pfs48/45 With Matrix-M Vaccine at Various Doses in Healthy Adult Volunteers by Assessing the Occurrence of Unsolicited Adverse Events (AEs) for 28 Days Following the Vaccination
Description: Number of unsolicited adverse events (AEs) for 28 days following the vaccination using e-diaries, clinical review, clinical examination (including observations) and laboratory results
Time Frame: 28 days following the vaccination
Population: A full list of unsolicited adverse events and the number of participants affected by each event is available in the 'Adverse events' section.
Measure: Number; unit: Number of events
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose
Number analyzed (Participants) | 8 | 8 | 1
Number of events
  Unsolicited adverse events - definitely related to the IMP | 0 | 0 | 1
  Unsolicited adverse events - probably related to the IMP | 7 | 3 | 0
  Unsolicited adverse events - possibly related to the IMP | 13 | 5 | 0
  Unsolicited adverse events - unlikely related to the IMP | 26 | 9 | 0
  Unsolicited adverse events - no relationship to the IMP | 8 | 6 | 0

4. Primary Outcome: Safety and Tolerability of the Pfs48/45 With Matrix-M Vaccine at Various Doses in Healthy Adult Volunteers. Assessed Through the Number of Participants With Abnormal Laboratory Test Results
Description: Occurrence of change from baseline laboratory tests
Time Frame: 28 days following vaccination
Measure: Number; unit: Number of participants with events
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose
Number analyzed (Participants) | 8 | 8 | 1
Number of participants with events
  Mild abnormalities | 5 | 4 | 0
  Moderate abnormalities | 0 | 1 | 0
  Severe abnormalities | 0 | 0 | 0

5. Primary Outcome: Safety and Tolerability of the Pfs48/45 With Matrix-M Vaccine at Various Doses in Healthy Adult Volunteers Assessed Through the Number of Participants With Serious Adverse Events
Description: Occurrence of serious adverse events will be presented according to local grading scales
Time Frame: Whole duration of the study (8 months following initial trial vaccination)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose
Number analyzed (Participants) | 8 | 8 | 1
Participants | 0 | 0 | 0

6. Primary Outcome: Safety and Tolerability of the Pfs48/45 With Matrix-M Vaccine at Various Doses in Healthy Adult Volunteers.
Description: Occurrence of AEs of special interest will be presented according to local grading scales and will be described in detail
Time Frame: Whole duration of the study (8 months following initial trial vaccination)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose
Number analyzed (Participants) | 8 | 8 | 1
Participants | 0 | 0 | 0

7. Secondary Outcome: Humoral Immunogenicity of the Pfs48/45 With Matrix-M Vaccine, When Administered to Healthy Adult Volunteers as Assessed by Humoral Responses to the Pfs48/45 Protein
Description: Antibody responses to the Pfs48/45 protein will be assessed through total IgG isotypes and avidity
Time Frame: Days 1, 29, 57, 140 and 240
Reporting Status: Not Posted

8. Secondary Outcome: Cellular Immunogenicity of the Pfs48/45 With Matrix-M Vaccine, When Administered to Healthy Adult Volunteers as Assessed by Cellular Responses to the Pfs48/45 Protein
Description: T cell responses to Pfs48/45 will be assessed by ex vivo enzyme-linked immunospot assays (ELISpot)
Time Frame: Days 1, 29, 57, 140 and 240
Reporting Status: Not Posted

9. Secondary Outcome: Ex Vivo Efficacy of the Pfs48/45 With Matrix-M Vaccine, When Administered to Healthy Adult Volunteers Using Direct Membrane Feeding Assays as Assessed by Transmission-reducing Activity
Description: Transmission-reducing activity
Time Frame: Days 1, 29, 57, 140 and 240
Reporting Status: Not Posted

10. Secondary Outcome: Ex Vivo Efficacy of the Pfs48/45 With Matrix-M Vaccine, When Administered to Healthy Adult Volunteers Using Direct Membrane Feeding Assays as Assessed by Transmission-blocking Activity
Description: Transmission-blocking activity
Time Frame: Days 1, 29, 57, 140 and 240
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrolment till the end of study visit for each volunteer (the duration of each volunteer's involvement in the study lasted up to 11.5 months).
Description: Systematic events collected via a participant-completed diary.
  Non-systematic events collected through a combination of the participant-completed diary and discussions at visits.
Arm/Group | Group 1 - Low Dose | Group 2 - Standard Dose | Group 3 - Fractional Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 7/8 | 7/8 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Low Dose (N=8) | Group 2 - Standard Dose (N=8) | Group 3 - Fractional Dose (N=1)
Nausea / Stomach issues (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) — Inc Acid Reflux, Gastrocolic, Gastroesophageal reflux, Stomach cramps
Back and shoulder ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bruising to vaccination site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) — inc: Dry Cough
covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dizzy spells (General disorders) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1) | 0 (0)
Headache (General disorders) | 7 (7) | 1 (1) | 0 (0)
Heavy feeling to arm of vaccination (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Infected Wisdom Tooth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injury to Coccyx (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Insect bites (General disorders) | 0 (0) | 1 (1) | 0 (0)
Itching to vaccination site (pruritus) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (General disorders) | 3 (4) | 1 (1) | 0 (0) — Inc Itchy Throat
Jaw Ache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Large Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhea/longer menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) — Inc: Longer menstrual bleeding, Period Pain
Migraine (Nervous system disorders) | 2 (9) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 0 (0) — Inc Runny Nose
Night Sweats (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nose Bleed (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pain at injection site (General disorders) | 1 (1) | 1 (1) | 0 (0) — These are the reports that were raised as AEs, as opposed to just being recorded on the participant diaries.
Pangs in hands (General disorders) | 1 (1) | 0 (0) | 0 (0)
Restlessness/insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Right upper limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Inc: Right Arm Pain, "Right Shoulder, Right Back and Right knee Pain"
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) — Inc Somnolence
Throat ulcers (General disorders) | 1 (1) | 0 (0) | 0 (0)
Tingling in left wrist (General disorders) | 1 (1) | 0 (0) | 0 (0)
Twisted ankle (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain at injection site - moderate (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 0 (0) — From participant diaries
Pain at injection site - mild (Skin and subcutaneous tissue disorders) | 7 (26) | 6 (25) | 0 (0) — From participant diaries
Itch at injection site - moderate (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) — From participant diaries
Itch at injection site - mild (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0) | 0 (0) — From participant diaries
Warmth at injection site - moderate (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — From participant diaries
Warmth at injection site - mild (Skin and subcutaneous tissue disorders) | 4 (9) | 6 (15) | 0 (0) — From participant diaries
Redness at injection site (Skin and subcutaneous tissue disorders) | 7 (76) | 5 (20) | 1 (1) — No redness was reported post Day7 after vaccination in participant diaries
Arthralgia - Moderate (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) — From participant diaries
Arthralgia - Mild (Musculoskeletal and connective tissue disorders) | 5 (9) | 3 (8) | 0 (0) — From participant diaries
Myalgia - Moderate (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) — From participant diaries
Myalgia - Mild (Musculoskeletal and connective tissue disorders) | 5 (13) | 5 (16) | 0 (0) — From participant diaries
Fever - Moderate (General disorders) | 3 (7) | 2 (2) | 0 (0) — From participant diaries
Fever - Mild (General disorders) | 2 (4) | 3 (4) | 0 (0) — From participant diaries
Headache - Moderate (General disorders) | 4 (5) | 4 (8) | 0 (0) — From participant diaries
Headache - Mild (General disorders) | 6 (47) | 7 (22) | 1 (2) — From participant diaries
Fatigue - Severe (General disorders) | 1 (1) | 0 (0) | 0 (0) — From participant diaries
Fatigue - Moderate (General disorders) | 2 (14) | 3 (3) | 0 (0) — From participant diaries
Fatigue - Mild (General disorders) | 6 (37) | 7 (20) | 0 (0) — From participant diaries
Nausea - Mild (General disorders) | 2 (2) | 3 (5) | 0 (0) — From participant diaries
Malaise - Moderate (General disorders) | 3 (6) | 1 (1) | 0 (0) — From participant diaries
Malaise - Mild (General disorders) | 5 (13) | 6 (14) | 0 (0) — From participant diaries

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT05400746/Prot_SAP_000.pdf